CLINICAL TRIAL: NCT06197204
Title: Biomarqueurs Diagnostiques, Pronostiques et de réponse au Traitement Dans l'Histiocytose Langerhansienne de l'Adulte
Brief Title: Biomarkers for Diagnostic, Prognostic and of Response to Treatment in Adult Langerhans Cell Histiocytosis
Acronym: BIOHISTIO
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230748
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Histiocytosis, Langerhans-Cell
MeSH Terms: conditions — Histiocytosis, Langerhans-Cell | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LCH patients
  Interventions: Other: Blood sampling; Other: Biopsy
- Control group: * diffuse lung cystic disease
  * pulmonary emphysema
  * healthy smokers
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — * at first visit in the reference center
  * at each follow-up visit ( once a year)
  * before and after specific treatment
  * in case of flare
  Groups: LCH patients
Other: Biopsy — In case of flare
  Groups: LCH patients
Other: Blood sampling — Once at inclusion visit
  Groups: Control group

SUMMARY:
Adult Langerhans histiocytosis (LCH) is a rare disease of unknown etiology, characterized by the activation of the MAPK (Mitogen-activated protein kinases) pathway, driven by various somatic mutations in the specific lesions of involved organs/tissues. LCH is currently classified as myeloid neoplasia with an inflammatory component. In patients with active systemic LCH, MAPK mutations may also be identified in plasma free cell DNA in patients. In contrast, circulating MAPK mutations seem more rarely detected in patients with LCH limited to a single organ/tissue (single system disease), but this has not been accurately assessed in a large series of patients.

The clinical presentation of LCH is very diverse, the prognosis variable, and the evolution marked by the occurrence of flares of the disease. A definitive diagnosis of LCH warrants histological confirmation obtained by a biopsy of an involved organ. In case of Pulmonary Langerhans cell histiocytosis (PLCH), a presumptive diagnosis is often acceptable when lung-computed tomography (CT) shows a nodulo-cystic pattern after excluding alternative diagnoses. In contrast, in case of purely cystic lung CT pattern, PLCH may be difficult to differentiate from other diffuse cystic lung diseases (mainly lymphangioléiomyomatose (LAM) and BHD (Birt-Hogg-Dubé syndrom), and eventually other rare disorders). Advanced PLCH may even be misdiagnosed as pulmonary emphysema that also occurs in smokers. In these situations, confirmation of PLCH warrants lung tissue, obtained most often by surgical lung biopsy that comprises significant morbidity or is not feasible in patients with altered lung function. Thus, the identification of specific blood biomarkers of cystic PLCH would be very useful.

On another hand, personalized management of adult patients with LCH is limited given the absence of predictive factors for prognosis or response to treatment.

The aim of this prospective study is to describe precisely the clinical phenotype at diagnosis and during follow-up of a large cohort of adult LCH patients and to seek for blood biomarkers eventually associated with prognosis or response to specific treatment. For patients with cystic PLCH specific markers for non-invasive diagnosis will also be investigated.

In the subgroup of patients with Single system (SS) LCH and specific driver MAPK mutation in tissue lesions, we will also look for the identification of this mutation in plasma free DNA at the time of a flare of the disease.

ELIGIBILITY:
Inclusion Criteria:

LCH patients :

* Age ≥ 18 years
* All confirmed LCH seen at the reference center whatever the clinical presentation

Controls :

* Age ≥ 18 years
* Patients with diffuse lung cystic disease, pulmonary emphysema and healthy smokers

All :

* Signing an informed consent
* Patients with health insurance

Exclusion Criteria:

* Persons under guardianship or curatorship, or deprived of freedom by a judicial or administrative decision.
* People benefiting from Medical Aid from the State (AME)
* Pregnant women, parturient and mothers who are breastfeeding.
* Persons subject to psychiatric care and persons admitted to a health or social establishment for purposes other than research
* Persons unable to express their consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult patients with LCH seen at the French reference center for histiocytoses.
  For the study on the diagnostic performance of blood biomarkers for cystic PLCH, a comparative group of patients with diffuse lung cystic diseases, pulmonary emphysema and healthy smokers will be included.
Sampling Method: Non-Probability Sample
Enrollment: 570 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2034-03-25 (Estimated); Study Completion 2034-03-25 (Estimated)

PRIMARY OUTCOMES:
Description of the clinical phenotype at diagnosis and the outcome of adult LCH patients | Up to 10 years

SECONDARY OUTCOMES:
Evaluation of the prognostic performance of blood biomarkers for adult LCH patients | Up to 10 years
Evaluation of the predictive performance of blood biomarkers for the therapeutic response | Up to 10 years
Evaluation of the diagnostic performance of blood biomarkers for patients with purely cystic Pulmonary Langerhans cell histiocytosis | Up to 10 years
Evaluation of the presence of MAPK tissue mutation in plasma cell free DNA for patients with Single System LCH at the time of a flare of the disease | Up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Louis, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided